CLINICAL TRIAL: NCT06257381
Title: Maximal Oxygen Uptake (VO2max) in Patients With COPD: a Test-Retest Reliability Study
Brief Title: Maximal Oxygen Uptake (VO2max) in Patients With COPD
Acronym: COPD-MAX
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Milan Mohammad, Medical student (BS.c.) at Department of Physical Activity Research Center, Rigshospitalet, Principal Investigator., Rigshospitalet, Denmark
Other Study IDs: H-23075064
Record Dates: First submitted 2024-02-05; First posted 2024-02-14 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: COPD
Keywords: Reliability; Test-retest; VO2max
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD-patients: We aim to include 16 patients with COPD across the FEV1% of predicted spectrum, ranging from mild to severe COPD. Participants will undergo lung function test and VO2max
  Interventions: Other: VO2max
- Matched healthy volunteers: We aim to include 16 healthy matched controls (sex +-3year age).
  Interventions: Other: VO2max

INTERVENTIONS:
Other: VO2max — Overall design 16 non-smoking individuals with COPD and 16 controls (non-smokers) matched for age and sex on a group level will be included in the study. The study consists of two study days. Separation between the study days are at least 48 hours and maximum 10 days.
  Before entering the study: Informed written and oral consent.
  Study day 1: Medical examination, full lung function testing (dynamic spirometry, whole-body plethysmography, diffusion capacity) followed by a maximal oxygen consumption test (VO2peak), VO2-verification bout and VO2kinetic test (duration 3h).
  Study day 2: Participants will undergo a maximal oxygen consumption test (VO2peak), VO2-verification bout and VO2kinetic test (duration 1,5h).
  Other Names: Lung function test

SUMMARY:
Patients with chronic obstructive pulmonary disease (COPD), facing a decline in lung function and compromised quality of life, often benefit from regular exercise (1). Assessing their cardiorespiratory fitness through maximal oxygen uptake (VO2max) is crucial (2), yet research on its validity and reliability in COPD patients remains sparse. This study aims to fill this gap, examining the content validity and test-retest reliability of the VO2-max test in COPD, comparing it with healthy controls.

DETAILED DESCRIPTION:
Introduction and background Patients with COPD face a challenging journey characterized by a progressive loss of lung function, ultimately resulting in a diminished quality of life, exercise limitations and heightened vulnerability to disability and premature mortality. Recognizing the pivotal role of regular exercise in enhancing the well-being of COPD patients, it becomes crucial to evaluate their cardiorespiratory fitness through parameters such as maximal oxygen uptake (VO2max). This metric serves as a cornerstone in assessing the maximal capacity of the cardiovascular system to deliver oxygen to working muscles and the muscles' ability to utilize oxygen during sustained exercise.

In broader health contexts high VO2max has been established as a key indicator inversely correlated with the risk of cardiovascular diseases and mortality. However, despite the acknowledged importance of VO2max, there is a notable gap in research focusing specifically on VO2max of COPD patients. The need for a thorough examination of the content validity of the VO2-max test in the context of COPD, along with an assessment of its test-retest reliability (day-to-day variation), has not been adequately addressed, especially in comparison with healthy individuals. While regular exercise has proven to be a transformative factor in improving the quality of life for COPD patients, there remains a critical need to explore the reliability of VO2-max testing within this population. Not only does COPD induce a decline in physical activity, but it can also contribute to a reduction in VO2-max. Consequently, understanding the validity and test-retest reliability of VO2-max testing in COPD becomes paramount.

Aim To compare the validity and test-retest reliability of the VO2-max test in COPD patients compared with healthy controls.

Perspective The results are relevant for designing future studies of VO2max and VO2kinetics as outcomes in COPD patients.

ELIGIBILITY:
Inclusion criteria - COPD patients

* Men and women
* 45-80 years
* COPD (GOLD stage I to IIII)
* Forced expiratory volume in 1 sec (FEV1)/forced vital capacity ratio (FVC) < 0.8, FEV1 < 90% of predicted value.
* Modified Medical Research Council score (mMRC 0 - 3)
* Resting arterial oxygenation > 90%

Inclusion criteria - healthy controls

* Men and women
* 45-80 years
* Normal FEV1, FVC, FEV1/FVC, and single-breath diffusion capacity
* Same sex, age (± 3 years) as the COPD patients

Exclusion criteria - COPD patients

* Symptoms of ischaemic heart disease
* Known heart failure
* Claudication
* Symptoms of disease within 2 weeks prior to the study
* Participation in pulmonary rehabilitation within 6 months
* Known malignant disease
* Pregnancy
* Unstable cardiac arrhythmic disease
* Renal or liver dysfunction

Exclusion criteria - healthy controls

* Known chronic lung disease
* Known ischaemic heart disease
* Known heart failure
* Symptoms of disease within 2 weeks prior to the study
* Known malignant disease
* Claudication
* Pregnancy
* Unstable cardiac arrhythmic disease
* Renal or liver dysfunction

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited through advertisements at pulmonary outpatient clinics and general practices in Greater Copenhagen, and by advertisements in newspapers, magazines, social media, and on forsøgsperson.dk as well as through forskningnu.dk. We have created a specific social media account which is used on different social medias to share knowledge and potentially recruit participants. It will not be possible to comment or tag people in our posts, and potentially interested participants will only be able to contact our research group via encrypted Region H mail. An e-mail address and telephone number will be provided by which interested participants can contact the research group.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Between-day smallest real difference (SRD) for VO2 peak in COPD vs. healthy controls | Measured at day 1 and day 2
Between-day coefficient of variance (CV) for VO2 peak in COPD vs. healthy controls (co-primary) | Measured at day 1 and day 2

SECONDARY OUTCOMES:
Between-day smallest real difference (SRD) Wmax in COPD vs. healthy controls | Measured at day 1 and day 2
Between-day coefficient of variance (CV) Wmax in COPD vs. healthy controls | Measured at day 1 and day 2
Between-day smallest real difference (SRD) RER at VO2 peak in COPD vs. healthy controls | Measured at day 1 and day 2
Between-day coefficient of variance (CV) RER at VO2 peak in COPD vs. healthy controls | Measured at day 1 and day 2
Between-day smallest real difference (SRD) Gas Exchange Threshold (GET) in COPD vs. healthy controls | Measured at day 1 and day 2
Between-day coefficient of variance (CV) Gas Exchange Threshold (GET) in COPD vs. healthy controls | Measured at day 1 and day 2
Between-day smallest real difference (SRD) in Ventilatory reserve in COPD vs. healthy controls | Measured at day 1 and day 2
Between-day coefficient of variance (CV) in Ventilatory reserve in COPD vs. healthy controls | Measured at day 1 and day 2
Between-day smallest real difference (SRD) and Between-day coefficient of variance (CV) in VE/VCO2 at GET in COPD vs. healthy controls | Measured at day 1 and day 2
Between-day smallest real difference (SRD) in VE/VCO2 at GET in COPD vs. healthy controls | Measured at day 1 and day 2
Between-day coefficient of variance (CV) in HR peak in COPD vs. healthy controls | Measured at day 1 and day 2

OTHER OUTCOMES:
End-expiratory lung volume at GET between-day smallest real difference (SRD) in COPD vs. healthy controls | Measured at day 1 and day 2
End-expiratory lung volume at GET between-day coefficient of variance (CV) in COPD vs. healthy controls | Measured at day 1 and day 2
End-expiratory lung volume at VO2peak between-day smallest real difference (SRD) in COPD vs. healthy controls | Measured at day 1 and day 2
End-expiratory lung volume at VO2peak between-day coefficient of variance (CV) in COPD vs. healthy controls | Measured at day 1 and day 2
Inspiratory capacity at GET between-day smallest real difference (SRD) in COPD vs. healthy controls | Measured at day 1 and day 2
Inspiratory capacity at GET between-day coefficient of variance (CV) in COPD vs. healthy controls | Measured at day 1 and day 2
Inspiratory capacity at VO2peak between-day smallest real difference (SRD) in COPD vs. healthy controls | Measured at day 1 and day 2
Inspiratory capacity at VO2peak between-day coefficient of variance (CV) in COPD vs. healthy controls | Measured at day 1 and day 2
Respiratory rate at GET between-day smallest real difference (SRD) in COPD vs. healthy controls | Measured at day 1 and day 2
Respiratory rate at GET between-day coefficient of variance (CV) in COPD vs. healthy controls | Measured at day 1 and day 2
Respiratory rate at VO2peak between-day smallest real difference (SRD) in COPD vs. healthy controls | Measured at day 1 and day 2
Respiratory rate at VO2peak between-day coefficient of variance (CV) in COPD vs. healthy controls | Measured at day 1 and day 2
Tidal volume at GET between-day smallest real difference (SRD) in COPD vs. healthy controls | Measured at day 1 and day 2
Tidal volume at GET between-day coefficient of variance (CV) in COPD vs. healthy controls | Measured at day 1 and day 2
Tidal volume at VO2peak between-day smallest real difference (SRD) in COPD vs. healthy controls | Measured at day 1 and day 2
Tidal volume at VO2peak between-day coefficient of variance (CV) in COPD vs. healthy controls | Measured at day 1 and day 2
Arterial saturation at GET between-day smallest real difference (SRD) in COPD vs. healthy controls | Measured at day 1 and day 2
Arterial saturation at GET between-day coefficient of variance (CV) in COPD vs. healthy controls | Measured at day 1 and day 2
Arterial saturation at VO2peak between-day smallest real difference (SRD) in COPD vs. healthy controls | Measured at day 1 and day 2
Arterial saturation at VO2peak between-day coefficient of variance (CV) in COPD vs. healthy controls | Measured at day 1 and day 2
Inspiratory time at GET between-day smallest real difference (SRD) in COPD vs. healthy controls | Measured at day 1 and day 2
Inspiratory time at GET between-day coefficient of variance (CV) in COPD vs. healthy controls | Measured at day 1 and day 2
Expiratory time at VO2peak between-day smallest real difference (SRD) in COPD vs. healthy controls | Measured at day 1 and day 2
Expiratory time at VO2peak between-day coefficient of variance (CV) in COPD vs. healthy controls | Measured at day 1 and day 2
Time constant (tau) from VO2 kinetic test between-day smallest real difference (SRD) in COPD vs. healthy controls | Measured at day 1 and day 2
Time constant (tau) from VO2 kinetic test between-day coefficient of variance (CV) in COPD vs. healthy controls | Measured at day 1 and day 2
Steady state gain from VO2 kinetic test between-day smallest real difference (SRD) in COPD vs. healthy controls | Measured at day 1 and day 2
Steady state gain from VO2 kinetic test between-day coefficient of variance (CV) in COPD vs. healthy controls | Measured at day 1 and day 2

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Aktiv Sundhed (CFAS), Rigshospitalet, Copenhagen, Denmark., Copenhagen, København Ø, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Will be decided upon study completion.